CLINICAL TRIAL: NCT05328310
Title: The Differential Effects of Antihypertensive Drugs on Central Blood Pressure: Comparison Between Beta-blocker and ARB
Brief Title: Effect of Different Antihypertensive Drugs on Central Blood Pressure
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Dr. Cheol Woong Yu, Clinical professor, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATD-CBP
Record Dates: First submitted 2022-02-08; First posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Nebivolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telmisartan (Active Comparator): Within enrolled patients who agreed to participate in the study, signed informed consent and being satisfied with inclusion and exclusion criteria, telmisartan is given as the primary antihypertensive agent.
  Interventions: Drug: Nebivolol
- Nebivolol (Experimental): Within enrolled patients who agreed to participate in the study, signed informed consent and being satisfied with inclusion and exclusion criteria, nebivolol is given as the primary antihypertensive agent.
  Interventions: Drug: Nebivolol

INTERVENTIONS:
Drug: Nebivolol — Treatment of nebivolol instead of telmisartan; the drug administration is mutually exclusive for the two arms.

SUMMARY:
Trial name) The differential effects of antihypertensive drugs on central blood pressure: comparison between beta-blocker(BB) and angiotensin receptor blocker ARB)

Objectives) To evaluate the effect of BB, which has vasodilatory effects, on CBP by comparison between ARB, one of the most widely used class of antihypertensives.

Study design) A multicenter, prospective, randomized, controlled, open-label clinical trial for hypertension patients.

Patient enrollment) 110 patients will be enrolled at 2 centers in South Korea.

Patient follow-up) Patients will go through an initial washout period of two weeks prior to randomization. After pre-medication baseline visit and randomization, clinical follow-up will occur at 4, 8, 12 weeks after initial administration of randomized drug. The follow-up visits are office visits.

Primary endpoint) Reduction in CBP at 12 weeks.

Secondary endpoints) Clinical events including adverse reactions to the drugs.

DETAILED DESCRIPTION:
1. Study background Different antihypertensive agents induce varied response in terms of CBP, even if peripheral BP-lowering effects are similar. In ASCOT-CAFE study, the atenolol±thiazide group and the amlodipine±perindopril group had similar efficacy in lowering peripheral BP, but CBP was significantly higher in the atenolol±thiazide group. This, amongst other studies, provided grounds for BBs being exempted from first-line therapy for hypertension.

   A possible explanation for this suboptimal performace of BB in lowering CBP is that in the atenolol±thiazide group, the lowered heart rate and subsequently an increase in systolic time promotes the augmentation of systolic pressure waves by the pressure wave reflections. Second, the comparatively high vasoconstricting effects of atenolol±thiazide group may result in a more proximal formation of pressure waves.

   Recently, third-generation BBs such as nebivolol have been developed, with additional vasodilatory effects which distinguishes them from previous BBs, and less accentuated heart rate-slowing effects. However, the effect of these new-generation of BBs on CBP is yet to be elucidated.
2. Study objectives The primary objective of this study is to evaluate the clinical efficacy of nebivolol, a BB, in lowering the CBP compared to telmisartan, an ARB.
3. Medical devices and therapeutic agents The medical devices and therapeutic agents to be used in this study are the treatment modalities that have been proven to be beneficial in the treatment of hypertensive patients without clear contraindications.
4. Expected effects of the research The clinical benefits of lowering CBP as well as peripherally measured BP have been previously described. Currently, the use of BBs in hypertensive patients is limited to those with clear indications such as concomitant atrial fibrillation or heart failure, due to its inferiority in lowering CBP compared to other antihypertensive agents. For those with coincident indications for BBs, or those with contraindications to other classes of antihypertensives, having a secure alternative first-line drug would be beneficial. This study is expected to give evidence for, or against, the use of BBs in hypertensive patients in terms of lowering the CBP in addition to PBP.
5. Clinical trial monitoring Monitor personnel designated by the investigator to obtain quality test data will review the clinical trial data at appropriate intervals to ensure accuracy, completeness, and compliance with the protocol. The monitoring personnel can investigate all documents and essential records held by clinical investigators or clinical trial laboratories, including the medical records (office, clinic, and hospital) of the subjects participating in the clinical trial. Clinical investigators and researchers should allow access to these records to the monitoring personnel. The monitoring plan will be conducted three times in total, at the time of registering the number of subjects corresponding to 50% or more of the total enrollment number, when the completed research subject reaches 70% or more, and immediately before the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. For patients with newly diagnosed hypertension: SBP ≥140mmHg or DBP ≥90 mmHg
2. For patients with prior diagnosis of hypertension: SBP ≥140mmHg or DBP ≥90 mmHg after a two-week washout period of previous antihypertensive medications.
3. Patients who wrote the informed consent: The subject should be able to receive informations of treatment, risks, effects and other therapeutic modalities regarding different antihypertensive agents at least verbally, and investigators should be provided written informed consent from a subject or a legally recognized representative prior to giving any treatment related to the study.

Exclusion Criteria:

1. Patients with contraindications or hypersensitive/allergic reactions to any class of antihypertensive agents.
2. Severe hypertension patients: SBP ≥200mmHg or DBP ≥110 mmHg at any visit during the study.
3. Chronic kidney disease (creatinine >1.5mg/dL)
4. Chronic obstructive pulmonary disease
5. Chronic heart failrue (LVEF ≤35%)
6. Patients who are pregnant or plan on becoming pregnant during the duration of the study, both male and female sex
7. Patients who are illiterate, have psychiatric illnesses or who do not agree to be enrolled in the study.
8. Other patients who are deemed unfit for the study as assessed by the investigators.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2019-01-06 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Central blood pressure | Initial admission date and follow-up visits at 4, 8, 12 weeks
  Differential changes in CBP by nebivolol and telmisartan

CONTACTS AND LOCATIONS:
Overall Officials: Cheol Woong Yu, M.D. Ph.D, Principal Investigator — Korea University Anam Hospital
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lim S, Kook H, Yu CW, Kim JH, Cha JJ, Joo HJ, Na JO, Choi CU, Lim SY, Park JH, Hong SJ, Lim DS. Differential Effects of Antihypertensive Drugs on Central Blood Pressure: A Randomized Comparison Between Nebivolol and Telmisartan. Am J Hypertens. 2026 Feb 1;39(2):303-311. doi: 10.1093/ajh/hpaf098. PMID 40490940